# **Cover Page**

### Official Title:

Assessing the Difference and Effectiveness of Art and Sandplay Therapy in Treating Posttraumatic Stress Disorders Among Syrian Refugee Children in Jordan

NCTXXXXXX (To be assigned upon registration)

Document Date: [Insert Date]

IRB Approval Number: 1/92/2014

Principal Investigators:
Dr. Abdallah Alzoubi
Dr. Khalid Ahmed Abdullah Kheirallah
Ms. Nour Khalid Bundogji

Funding Source:

Faculty Member Research Grant (FMRG), Jordan University of Science and Technology

Ethical Approval Date:

Approved by the Institutional Research Board (IRB) on December 16, 2014

## 1. Executive Summary

This study aims to evaluate the effectiveness of art therapy and sandplay therapy in reducing symptoms of Posttraumatic Stress Disorder (PTSD) among Syrian refugee children aged 6–12 living in Jordan. The study employs a randomized controlled trial (RCT) design with three groups: sandplay therapy, art therapy, and a control group. Participants will undergo 12 weeks of intervention, with pre- and post-intervention assessments using the Harvard Trauma Questionnaire (HTQ). The study has received ethical approval from the Institutional Research Board (IRB) of Jordan University of Science and Technology (Approval No. GM7601).

## 2. Background and Rationale

Posttraumatic stress disorder (PTSD) is a significant mental health concern among refugee children exposed to war-related trauma. Traditional treatments such as Eye Movement Desensitization and Reprocessing (EMDR) and Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) are effective but may not benefit all patients, particularly those with poor verbal memory or prolonged trauma exposure. Nonverbal therapies like sandplay and art therapy offer alternative approaches that may be more accessible and culturally sensitive for refugee populations. This study seeks to provide evidence for the clinical use of these therapies in treating PTSD among Syrian refugee children.

## 3. Study Objectives

- 1. To determine the difference in effectiveness between art therapy and sandplay therapy compared to each other and to a control group.
- 2. To evaluate whether sandplay therapy results in greater improvement in PTSD symptoms compared to art therapy.

### 4. Study Design and Methodology

### **Study Population**

- Target Population: Syrian refugee children aged 6–12 living in Jordan.
- Sample Size: 90 children (30 per group: sandplay, art therapy, control).

#### **Inclusion Criteria**

- Diagnosed with PTSD related to war trauma (e.g., witnessed death, shrapnel injuries, war violence).
- Aged 6-12 years.
- Residing in Jordan as refugees due to the Syrian Civil War.

#### **Exclusion Criteria**

- Pre-existing psychosocial issues unrelated to war trauma.

## **Randomization and Group Allocation**

Participants will be randomly assigned to one of three groups:

- 1. Sandplay therapy group.
- 2. Art therapy group.
- 3. Control group (no formal therapy).

#### Interventions

- Sandplay Therapy: Participants will create scenes in a sandbox using miniature objects. Sessions last 20–30 minutes.
- Art Therapy: Participants will draw using coloring utensils on blank paper. Sessions last 30 minutes.
- Control Group: No formal therapy.

#### **Outcome Measures**

Primary outcome: Change in PTSD severity scores measured using the Harvard Trauma Questionnaire (HTQ). Scores will be categorized as mild, moderate, or severe based on a 16-item scale rated 1–4.

#### Location

Zad Children Center, Amman, Jordan.

## **Duration**

- Total duration: 14 weeks.
- Intervention period: 12 weeks.
- Pre- and post-assessment sessions: Weeks 1 and 14.

### **Session Details**

- Session 1: Establish rapport, obtain consent, and conduct pre-assessment.
- Sessions 2–13: Weekly therapy sessions for sandplay and art therapy groups.
- Session 14: Post-assessment and closing meeting.

### **Data Collection**

- HTQ administered at baseline and post-intervention.
- Photographs of sandplay creations and art pieces for documentation.

## 6. Statistical Analysis Plan

### **Primary Analysis**

- Paired t-test: Compare pre- and post-intervention mean scores within each group.
- Independent t-test: Compare mean differences between groups (sandplay vs. art therapy, sandplay vs. control, art therapy vs. control).

# **Secondary Analysis**

- Subgroup analysis by age and gender.
- Correlation analysis between session attendance and symptom improvement.

# Significance Level

p-value < 0.05 will be considered statistically significant.

### 7. Ethical Considerations

- Informed Consent: Obtained from legal guardians of all participants.
- Confidentiality: Participant data will remain anonymous.
- Withdrawal Rights: Participants can withdraw from the study at any time without penalty.
- Safety Measures: Therapists will ensure a safe and supportive environment during sessions.
- IRB was secured from King Abdulla University Teaching Hospital in Irbid, Jordan.

## 8. References

- 1. American Psychiatric Association. (2000). Diagnostic and statistical manual of mental disorders (4th ed., Text Revision).
- 2. Bisson, J. I., Ehlers, A., Matthews, R., Pilling, S., Richards, D., & Turner, S. (2007). Psychological treatments for chronic post-traumatic stress disorder: Systematic review and meta-analysis. \*British Journal of Psychiatry\*, 190, 97–104. PMID: 17290083
- 3. Schoumen, T., et al. (2014). Art therapy and sandplay therapy in PTSD treatment.
- 4. Harvard Trauma Questionnaire (HTQ). (2011). Harvard Program in Refugee Trauma.